CLINICAL TRIAL: NCT04536428
Title: ClearEndoclip Versus EZ Clip for the Hemostasis of Upper Gastrointestinal Ulcer Bleeding: an Open-label, Non-inferiority, Randomized, Multicenter Trial
Brief Title: ClearEndoclip Versus EZ Clip for Upper Gastrointestinal Ulcer Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); National Cancer Center, Korea (Other Government); Nowon Eulji Medical Center (Unknown); Pusan National University Hospital (Other); Wonju Severance Christian Hospital (Other); Inha University Hospital (Other); Presbyterian medical center (Unknown)
Responsible Party: Principal Investigator, Sun Gyo Lim, MD, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-DEV-DE2-20-148
Record Dates: First submitted 2020-08-06; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: peptic ulcer; hemorrhage; stomach; duodenum
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Peptic Ulcer; Hemorrhage | interventions — Hemostasis, Endoscopic; Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ClearEndoclip (Experimental): This arm is a group in whom ClearEndoclip would be used for the treatment of bleeding.
  Interventions: Device: Endoscopic hemostasis with clip
- EZ clip (Active Comparator): This arm is a group in whom EZ clip would be used for the treatment of bleeding.
  Interventions: Device: Endoscopic hemostasis with clip

INTERVENTIONS:
Device: Endoscopic hemostasis with clip — This intervention is performed as the following orders.
  * The tip of endoscope is accessed to a bleeding site.
  * The accurate visualization of bleeding site is done.
  * A sheath of delivery system of clip is inserted through a working channel of endoscope.
  * The end of clip is opened in front of the bleeding site. If needed, clip could be rotated to adjust to a bleeding target.
  * The both ends of clip are placed on both sides of a bleeding site.
  * If bleeding is still continued, additional placements of clip are tried until bleeding stops.

SUMMARY:
We are going to conduct a comparative study to analyze the clinical effectiveness and user convenience of EZ clips that have been used in upper gastrointestinal ulcer bleeding and newly developed clip (ClearEndoclip, FineMedix, Taegu) in Korea.

1) Research hypothesis and purpose

* This study was designed to prove the hypothesis that the hemostatic effect of newly developed endoscopic clip (ClearEndoclip, FineMedix, Taegu, Korea) is not inferior to that of EZ clip (Olympus, Tokyo, Japan) in the treatment of hemostasis for patients who visited the upper gastrointestinal ulcer bleeding.
* This study was designed as a multi-center (9 institutions), open-labelled, randomized comparative clinical trial (1:1 ratio).

DETAILED DESCRIPTION:
1. Design of this study

   1. Stratified randomization is performed, and the variable used for stratification is the patient's age (65 years or older, 65 years or less).
   2. The existing clip (control) and the domestic clip (experimental group) are divided by the block size randomization method of size 4 for each floor.
2. Patients and Methods

   1. inclusion criteria

      * Men and women aged 20 to 80
      * The patients who came to the emergency room due to upper gastrointestinal bleeding with as follows: peptic ulcer with acute bleeding or protruding vascular exposure (Forrest class Ia-IIa), anastomotic vascular ulcer bleeding, bleeding from endoscopic submucosal dissection or endoscopic mucosal resection site after 24 hours
      * American Society of Anesthesiologist (ASA) Physical Status 1 - 3
      * Patients with adequate patient compliance and adequate geographical distance for follow-up. character
   2. exclusion criteria

      * Patients with gastrointestinal bleeding who are not recommended to clip Bleeding from a malignant tumor Hemorrhagic gastritis Angiodysplasia variceal bleeding
      * Bleeding during endoscopic submucosal dissection or endoscopic mucosal resection
      * Patients with insufficient clinical information
      * Pregnant or lactating patients
      * Patients or guardians who have not obtained informed consent
   3. The number of patients

      * The number of subjects was calculated based on a non-inferiority study

        * The reported rate of rebleeding after hemostasis using the conventional hemoclip: about 5%.
        * 2.5% one-sided test, 80% power, and non-inferiority limit set to 10%

          * 75 subjects are required for each group, and 83 subjects are required if the drop rate is assumed to be 10%.
   4. Methods

      * After completing an informed consent form to the subjects who wish to participate in the study at the time of visit, basic clinical variables are checked.
      * First endoscopic hemostasis is performed. In this time, EZ clip is used for the subjects assigned to the control group, and ClearEndoclip is used for the subjects assigned to the experimental group to target blood vessels in the ulcer. At the same time, clinical parameters related to hemostasis are recorded.
      * After hemostasis is performed, rebleeding and complications are tracked up to 30 days after the procedure.
   5. Variables to be collected

      * At the time of visit: age, gender, height, weight, drug use (anticoagulant/antiplatelet agents, NSAIDs, steroids), underlying diseases (cirrhosis, diabetes, end-stage renal failure, heart disease, lung disease), hematological data, hemoglobin, Complete Rockall score
      * At the time of primary endoscopic hemostasis: location of ulcer, size of ulcer, size of exposed blood vessel (based on 2mm), forrest classification, total number of clips used, number of failed clips, usage and usage of epinephrine, procedure time (minutes) , Clip hemostasis success, treatment after clip hemostasis failure
      * After hemostasis: rebleeding (within 7 days), number of clips and bleeding from the follow-up endoscope after 48 hours, death within 30 days, ICU hospitalization date, total hospitalization date, complications of hemostasis, Helicobacter pylori

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 to 80
* The patients who came to the emergency room due to upper gastrointestinal bleeding with as follows: peptic ulcer with acute bleeding or protruding vascular exposure (Forrest class Ia-IIa), anastomotic vascular ulcer bleeding, bleeding from endoscopic submucosal dissection or endoscopic mucosal resection site after 24 hours
* American Society of Anesthesiologist (ASA) Physical Status 1 - 3
* Patients with adequate patient compliance and adequate geographical distance for follow-up. character

Exclusion Criteria:

* Patients with gastrointestinal bleeding who are not recommended to clip Bleeding from a malignant tumor Hemorrhagic gastritis Angiodysplasia variceal bleeding
* Bleeding during endoscopic submucosal dissection or endoscopic mucosal resection
* Patients with insufficient clinical information
* Pregnant or lactating patients
* Patients or guardians who have not obtained informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate after endoscopic hemostasis | upto 7 days
  The rate of rebleeding at the site of bleeding within 7 days after the first endoscopic hemostasis, which should be identified endoscopically.

SECONDARY OUTCOMES:
Satisfaction scores of the operator and the assistant | during endoscopic procedure
  the degree in ten-scale in terms of an endoscopic visibility to a bleeding site and the easiness of use. the minimum: 1(worst value), the maximum: 10(best)
Failure rate of clip installation | during endoscopic procedure
  Ratio of unsuccessful clips to total number of clips used

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gyo Lim, Principal Investigator — Department of Gastroenterology, Ajou University School of Medicine
Locations (1):
- Sun Gyo Lim, Suwon, Gyeonggi-do, South Korea